CLINICAL TRIAL: NCT00004585
Title: A Phase IV, Open-Label, Multicenter Study of the Efficacy and Safety of Quadruple Combination Antiretroviral Therapy With Combivir (Lamivudine 150mg/Zidovudine 300mg) BID, Ziagen (Abacavir) 300mg BID, and Sustiva (Efavirenz) 600mg QD for 24 Weeks, Followed by the Triple Nucleoside Combination Tablet (Abacavir 300mg/Lamivudine 150mg/Zidovudine 300mg) BID Plus Sustiva (Efavirenz) 600mg QD for 24 Weeks in HIV-Infected Adults
Brief Title: A Study of the Safety and Effectiveness of Combination Anti-HIV Therapy in HIV-Infected Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 307A; COL30336
Record Dates: First submitted 2000-02-15; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-11

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Zidovudine; Lamivudine; RNA, Viral; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; abacavir; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — abacavir; Lamivudine; Zidovudine; lamivudine, zidovudine drug combination; efavirenz

INTERVENTIONS:
Drug: Abacavir sulfate, Lamivudine and Zidovudine
Drug: Lamivudine/Zidovudine
Drug: Abacavir sulfate
Drug: Efavirenz

SUMMARY:
The purpose of this study is to see if a certain combination of anti-HIV drugs is safe and effective in HIV-infected patients. The drug combination includes a tablet containing lamivudine and zidovudine (called Combivir) plus abacavir plus efavirenz.

DETAILED DESCRIPTION:
Patients take open-label Combivir plus abacavir plus efavirenz for 48 weeks. [AS PER AMENDMENT 4/20/00: Patients taking Combivir plus abacavir at Week 24 receive the triple-nucleoside-combination tablet (TCT) (abacavir/lamivudine/zidovudine) beginning at Week 24 and continuing through Week 48, in combination with efavirenz (or nevirapine if the patient has made a protocol-allowed substitution). Patients not taking Combivir and abacavir at Week 24 will continue in the study on the substituted protocol-allowed drug regimen, provided their plasma HIV RNA is below 400 copies/ml at 24 weeks.] Following enrollment on Study Day 1, on-study evaluations (virologic and safety) are performed at Weeks 2, 4, 8, 12, 16, and then every 8 weeks through Week 48 (end of study). CD4 evaluations are performed at baseline and at Weeks 4, 8, and then every 8 weeks through Week 48. Immune reconstitution testing is performed at baseline and at Weeks 12, 24, and 48. Patients complete the PMAQ7 version 1.1 medication adherence questionnaire at Weeks 2, 8, 12, 24, and 48 (or at their last study visit). All patients are requested to return for a post-study follow-up evaluation 2 to 4 weeks after the last on-study visit. Patients must have a plasma HIV RNA less than 400 copies/ml at Week 24 in order to continue in the study.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have HIV levels of 50,000 copies/ml or more within 21 days prior to starting treatment.
* Are at least 18 years of age.
* Are willing to use an effective method of birth control during the study.
* (This study has been changed. A CD4 cell count of 50/mm3 or more within 21 days prior to starting treatment is no longer required.)

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are pregnant.
* Have AIDS.
* Cannot take medications by mouth.
* Have hepatitis and it is active.
* Are enrolled in other investigational drug studies.
* Are allergic to any of the study drugs.
* Have a serious medical condition, such as heart disease.
* Have ever taken certain anti-HIV drugs such as nonnucleoside reverse transcriptase inhibitors (NNRTIs) or protease inhibitors (PIs).
* Have ever had more than 7 days of treatment with a nucleoside reverse transcriptase inhibitor (NRTI). Patients should have no prior treatment with abacavir and no prior treatment with at least one of the following: lamivudine or zidovudine.
* Have had radiation therapy or chemotherapy within 4 weeks prior to study entry, or plan to have such therapy during the study.
* Have received medications that might affect the immune system, such as systemic corticosteroids, interleukins, vaccines, or interferons within 4 weeks prior to study entry.
* Have received an HIV vaccine within 3 months prior to study entry.
* Are taking foscarnet, hydroxyurea, or other drugs that work against HIV.
* Have taken certain medications such as astemizole, cisapride, dihydroergotamine, ergotamine, ganciclovir, interferon-alpha, midazolam, terfenadine, and triazolam within 21 days of study entry.
* Abuse alcohol or drugs.
* Are unable to complete the whole study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 1999-10

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Tower Infectious Diseases / Med Associates Inc, Los Angeles, California
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - North Shore Univ Hosp, Manhasset, New York
  - Thomas Jefferson Univ, Philadelphia, Pennsylvania
  - Dallas Veterans Administration Med Ctr, Dallas, Texas